CLINICAL TRIAL: NCT07294001
Title: A Pilot Randomized Controlled Trial Of Shame-Focused Cognitive Behavioral Therapy For Suicide Prevention In Adolescent Psychiatric Inpatients
Brief Title: Shame-Focused Cognitive Behavioral Therapy For Reducing Suicide Risk In Adolescent Psychiatric Inpatients (SF-CBT)
Acronym: SF-CBT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University (Other)
Collaborators: Peking University Sixth Hospital (Other)
Responsible Party: Principal Investigator, Yinyin Zang, PhD, Principle Investigator, Peking University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SF-CBT-YouthSuicide-2025; IRB Approval No. 2025-69 (Other: Peking University Sixth Hospital Ethics Committee)
Record Dates: First submitted 2025-11-17; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-11

CONDITIONS: Adolescent Suicide; Suicidal Ideation; Suicidal Behavior; Shame
Keywords: Adolescents; Suicide Prevention; Suicidal Ideation; Suicidal Behavior; Shame; Cognitive Behavioral Therapy (CBT); Shame-Focused Cognitive Behavioral Therapy (SF-CBT); Randomized Controlled Trial (RCT); Feasibility Study; Pilot Trial; Psychiatric Inpatient
MeSH Terms: conditions — Suicidal Ideation; Suicide Prevention | interventions — Palliative Care

STUDY DESIGN:
Intervention Model Description: This is a randomized, parallel-group pilot trial. Participants will be allocated in a 2:1 ratio to receive either Shame-Focused Cognitive Behavioral Therapy (SF-CBT) plus parent sessions or supportive therapy plus parent sessions. Both groups will undergo 7 individual sessions and 3 parent sessions during hospitalization, followed by follow-up assessments at 1, 3, and 6 months.
Who Masked: Outcomes Assessor
Masking Description: This study uses a single-blind design. Only the independent outcomes assessors are masked to treatment allocation. Participants, care providers, and investigators are aware of group assignments due to the nature of the intervention. Outcome assessors remain blinded throughout baseline, post-treatment, and follow-up assessments to minimize bias.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Shame-Focused Cognitive Behavioral Therapy (SF-CBT) (Experimental): Participants in this arm will receive Shame-Focused Cognitive Behavioral Therapy (SF-CBT), a structured individual intervention targeting maladaptive shame coping patterns. The intervention consists of 7 individual sessions (50-60 minutes each), focusing on motivation building, emotion identification, behavioral chain analysis, cognitive restructuring of shame-related self-criticism and withdrawal, development of healthy self-esteem, and relapse prevention. Additionally, caregivers will participate in 3 psychoeducation sessions covering empathic communication, crisis management, and boundary setting, supported by AI-based scenario practice.
  Interventions: Behavioral: Shame-Focused Cognitive Behavioral Therapy (SF-CBT)
- Active Comparator: Supportive Therapy (ST) (Active Comparator): Participants in this arm will receive Supportive Therapy (ST), which emphasizes emotional support, therapeutic alliance, and adjustment to hospitalization. The intervention includes 7 individual sessions (50-60 minutes each) focusing on relationship building, emotional expression, and support for daily coping. Caregivers in this arm will also attend 3 psychoeducation sessions identical to those provided in the experimental group, covering empathic communication, crisis management, and boundary management.
  Interventions: Behavioral: Supportive Therapy (ST)

INTERVENTIONS:
Behavioral: Shame-Focused Cognitive Behavioral Therapy (SF-CBT) — A structured, manualized individual psychotherapy program consisting of 7 sessions (50-60 minutes each), delivered during hospitalization. The intervention includes modules on motivation building, emotional recognition, behavior chain analysis, shame coping strategies, self-esteem enhancement, and relapse prevention. In addition, caregivers participate in 3 psychoeducation sessions covering empathic communication, crisis response, and boundary management, supplemented by AI-assisted scenario simulations.
  Arms: Experimental: Shame-Focused Cognitive Behavioral Therapy (SF-CBT)
Behavioral: Supportive Therapy (ST) — A supportive counseling program consisting of 7 sessions (50-60 minutes each), focusing on relationship building, emotional support, and adaptation to hospitalization. Caregivers in this arm also receive 3 psychoeducation sessions identical to those in the experimental arm, covering communication, crisis management, and boundary setting, with AI-assisted practice.
  Arms: Active Comparator: Supportive Therapy (ST)

SUMMARY:
This pilot randomized controlled trial (RCT) aims to evaluate the feasibility, acceptability, and preliminary efficacy of Shame-Focused Cognitive Behavioral Therapy (SF-CBT) among high-risk psychiatric inpatient adolescents. Shame has been identified as a critical psychological mechanism underlying suicidal ideation and behavior, yet few interventions directly target it. SF-CBT is a structured, manualized intervention designed to reduce shame, improve coping strategies, and lower suicide risk.

Approximately 42 adolescents aged 13-18 years, admitted for recent suicide attempt or severe suicidal ideation, will be randomized in a 2:1 ratio to receive either SF-CBT or supportive therapy (ST). Both conditions include 7 individual sessions for adolescents and 3 structured psychoeducation sessions for parents/guardians.

Primary outcomes include feasibility metrics (recruitment, retention, adherence, fidelity, adverse events) and acceptability ratings from adolescents, parents, and therapists. Secondary outcomes include changes in suicidal ideation, suicidal behavior, shame, and coping styles, assessed at baseline, post-treatment, and 1-, 3-, and 6-month follow-ups.

Findings will inform refinement of the intervention manual, establish feasibility benchmarks, and provide effect size estimates to guide a subsequent large-scale RCT.

DETAILED DESCRIPTION:
Adolescent suicide is a major public health concern in China and worldwide. Shame, a powerful and often overlooked psychological driver of suicide risk, has rarely been the focus of intervention efforts. This study introduces and tests Shame-Focused Cognitive Behavioral Therapy (SF-CBT), a manualized and structured therapy designed specifically to reduce shame, enhance adaptive coping, and mitigate suicide risk in high-risk inpatient adolescents.

Objectives The primary objective is to test the feasibility and acceptability of SF-CBT in an inpatient psychiatric setting. Secondary objectives are to explore its preliminary efficacy in reducing shame, suicidal ideation, and suicidal behavior, and to evaluate the maintenance of effects at 1-, 3-, and 6-month follow-ups.

Design and Participants This is a single-site, single-blind pilot RCT conducted at Peking University Sixth Hospital adolescent psychiatric ward. Forty-two adolescents (ages 13-18) admitted with recent suicidal ideation or attempt and elevated baseline shame will be recruited. Exclusion criteria include acute mania, psychotic disorders, severe cognitive impairment, or expected hospitalization shorter than 14 days. Eligible participants will be randomized (2:1) to SF-CBT (~28) or ST (~14).

Intervention

SF-CBT: Seven 50-60 minute individual sessions covering motivation building, emotion recognition and chain analysis, shame-coping strategies, self-esteem enhancement, and relapse prevention. Parents/guardians will attend 3 psychoeducation sessions on empathic communication, crisis management, and family boundary-setting, supported by AI-based scenario simulations.

Supportive Therapy (ST): Seven supportive counseling sessions focusing on emotional support and inpatient adjustment. Parent psychoeducation sessions identical to SF-CBT arm.

Outcomes

Primary outcomes: Feasibility (recruitment and retention rates, adherence, fidelity, adverse events) and acceptability (satisfaction ratings by adolescents, parents, therapists).

Secondary outcomes: Suicidal ideation and behavior (C-SSRS, SIQ), shame (EISS), and shame-coping (CoSS), assessed at baseline, post-treatment, and 1-, 3-, and 6-month follow-ups.

Analysis and Significance Feasibility benchmarks (e.g., ≥70% recruitment, ≥80% completion) will guide readiness for a full-scale RCT. Preliminary efficacy will be explored using multilevel models, with effect sizes reported to inform sample size estimation.

This pilot study will establish the feasibility and safety of SF-CBT in high-risk adolescent inpatients and provide initial evidence for its impact on shame and suicide risk. Results will directly inform a larger RCT and contribute to evidence-based, mechanism-driven suicide prevention strategies for adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents aged 13-18 years, male or female.
* Recent suicide risk, defined as:

At least one suicide attempt in the past month, or Current suicidal ideation within the past month (with or without plan/intent) and at least one previous attempt.

* Elevated shame level (baseline score ≥ 9 on the External and Internal Shame Scale, EISS).
* Adequate cognitive capacity to participate in interviews and assessments.
* Parent/legal guardian (or designated responsible adult authorized by guardian) provides informed consent and agrees to participate.

Exclusion Criteria:

* Current manic episode.
* History of schizophrenia spectrum disorder, intellectual disability, or organic brain disease.
* Severe psychiatric or medical conditions that impair capacity for consent or participation.
* Expected to receive electroconvulsive therapy (ECT) during hospitalization.
* Anticipated inpatient stay shorter than 14 days (to ensure intervention completion).

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-08-10 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
The Columbia-Suicide Severity Rating Scale (C-SSRS) | Time Frame: Baseline, Week 4, Month 2, Month 5, and Month 7
  It will be used to assess suicidal ideation and suicidal behaviors (Posner et al., 2011). The C-SSRS is widely utilized in suicide risk assessment. It evaluates several aspects, including the presence of a suicide attempt, an interrupted attempt (prevented by external factors), an aborted attempt (self-terminated by the individual), preparatory or related suicidal behaviors, and lethality ratings.
  The actual lethality is rated on a 6-point scale. The potential lethality is rated on a 3-point scale (if actual lethality = 0), where 0 = "behavior unlikely to result in injury," and 2 = "likely to result in death even with medical intervention." Additionally, the presence of non-suicidal self-injury (NSSI) will be assessed, as it is associated with future suicide attempt risk. it is highly sensitive in detecting changes in suicidal behavior during treatment and can predict future suicidal behaviors and readmission(Ji et al., 2023).
The Columbia-Suicide Severity Rating Scale (C-SSRS) | Time Frame: Baseline, Week 4, Month 2, Month 5, and Month 7
  The C-SSRS will also be used to evaluate suicidal ideation and intent, with assessment time points identical to those above. Two subscales will be extracted for this study:
  Severity: Scores range from 1 to 5, representing "wish to be dead," "non-specific active suicidal thoughts," "suicidal thoughts with method," "suicidal intent," and "suicidal intent with a specific plan," respectively.
  Intensity: Evaluates the frequency, duration, controllability, deterrents, and reasons for suicidal ideation.

SECONDARY OUTCOMES:
The External and Internal Shame Scale, EISS | Baseline, Week 4, Month 2, Month 5, and Month 7
  Shame will be measured using the External and Internal Shame Scale (EISS), which assesses two core dimensions of shame as a transdiagnostic emotion: external shame and internal shame. Both the subscales and total scores of the EISS demonstrate good internal consistency and concurrent validity and are significantly associated with depressive symptoms (Ferreira et al., 2022).
The Compass of Shame Scale (CoSS) | Baseline, Week 4, Month 2, Month 5, and Month 7
  Coping or defensive strategies toward shame have a significant impact on psychological functioning. The Compass of Shame Scale (CoSS) will be used to assess four coping styles individuals employ when experiencing shame: attack self, withdrawal, attack others, and avoidance. Studies have shown that the CoSS has good reliability and validity, with internal consistency coefficients ranging from 0.74 to 0.91 across subscales (Elison et al., 2006).
The Alexian Brothers Urge to Self-Injure Scale (ABUSI) | Baseline, Week 4, Month 2, Month 5, and Month 7
  The Alexian Brothers Urge to Self-Injure Scale (ABUSI), which measures the severity of urges to engage in NSSI. The ABUSI shows good internal consistency, test-retest reliability, sensitivity to change, as well as convergent, predictive, and incremental validity (Washburn et al., 2010).
Deliberate Self-Harm Inventory (DSHI) | Baseline, Week 4, Month 2, Month 5, and Month 7
  The Deliberate Self-Harm Inventory (DSHI), which assesses deliberate self-harming behaviors. The DSHI demonstrates high internal consistency and good structural, convergent, discriminant, and test-retest validity, supporting its reliability and validity as a measure of deliberate self-harm (Gratz, 2001).
Patient Health Questionnaire-9, PHQ-9 | Baseline, Week 4, Month 2, Month 5, and Month 7
  Depression will be assessed using the Patient Health Questionnaire-9 (PHQ-9) (Kroenke et al., 2001). A study of 10,933 school-aged adolescents in Hong Kong found that the PHQ-9 demonstrated good model fit under a single-factor model with correlated item pairs and maintained measurement invariance across gender and age groups. The PHQ-9 exhibited good internal consistency (>0.84) and showed expected correlations with anxiety (>0.77), self-esteem (<-0.57), and perceived control (<-0.56). Therefore, the PHQ-9 is suitable for assessing and comparing depression severity among adolescents of different genders and age groups (Leung et al., 2020).
The Generalized Anxiety Disorder-7 (GAD-7) | Baseline, Week 4, Month 2, Month 5, and Month 7
  The Generalized Anxiety Disorder-7 (GAD-7) scale will be used to assess the severity of generalized anxiety disorder (GAD) symptoms. Research indicates that the GAD-7 has good internal consistency and demonstrates strong convergent validity with measures of anxiety, worry, depression, and stress. Moreover, the scale is highly sensitive to symptom changes during brief intensive cognitive-behavioral therapy (CBT). Overall, the GAD-7 shows excellent internal consistency, convergent validity, and sensitivity to change within this sample (Kertz et al., 2013).
Emotional Awareness Questionnaire, EAQ | Baseline, Week 4, Month 2, Month 5, and Month 7
  The Chinese version of the Insomnia Severity Index (ISI-C) will be used to evaluate the severity of insomnia in clinical patients. Studies have shown that the ISI-C has good reliability and validity, with a Cronbach's α of 0.804 and a test-retest reliability of 0.887 (P < 0.01). It also demonstrates good structural and predictive validity. When the cutoff score is set at 10.5, the ISI-C achieves 84.0% sensitivity and 92.3% specificity (P < 0.01) (Bai et al., 2018).
A self-developed Adolescent Irritability Scale | Baseline, Week 4, Month 2, Month 5, and Month 7
  A self-developed Adolescent Irritability Scale will be used, comprising four dimensions: self-injurious irritability, object-destructive irritability, interpersonal irritability, and self-directed irritability. Preliminary results indicate that the scale has good reliability and validity, and related psychometric research is currently in publication.
Rosenberg Positive Self-Esteem Scale, RSES | Baseline, Week 4, Month 2, Month 5, and Month 7
  The Chinese version of the Rosenberg Positive Self-Esteem Scale (RSES) will be used to measure levels of self-esteem. The RSES shows good item discrimination across different samples. Internal consistency reliability (Cronbach's α) ranges from 0.83 to 0.89 in college, adult, and military samples, while the four-week test-retest reliability in high school students is 0.76, indicating good structural validity (Chen et al., 2015).
Instability of Self-Esteem Scale, ISES | Baseline, Week 4, Month 2, Month 5, and Month 7
  The Instability of Self-Esteem Scale (ISES) will be used to evaluate fluctuations in self-esteem levels. Findings suggest that the ISES has satisfactory internal consistency and test-retest reliability. Moreover, its low correlation with the RSES indicates that the two instruments measure relatively independent psychological constructs. Distinct correlation patterns between ISES, CES-D, and BPI further support its discriminant validity (Chabrol et al., 2006).
The Self-Compassion Scale-Youth Version (SCS-Y) | Baseline, Week 4, Month 2, Month 5, and Month 7
  The Self-Compassion Scale-Youth Version (SCS-Y) will be used to assess self-compassion among early adolescents. It consists of six dimensions: self-kindness, self-judgment, mindfulness, isolation, common humanity, and over-identification. The SCS-Y demonstrates good test-retest reliability and construct validity, with expected correlations with mindfulness, well-being, life satisfaction, depression, psychological resilience, and achievement goal orientation (Neff et al., 2021).
The 2-Way Social Support Scale (2-Way SSS) | Baseline, Week 4, Month 2, Month 5, and Month 7
  The 2-Way Social Support Scale (2-Way SSS) will be used to evaluate both the giving and receiving of social support, distinguishing two primary types: emotional support and instrumental support. It consists of four core dimensions: (a) giving emotional support, (b) giving instrumental support, (c) receiving emotional support, and (d) receiving instrumental support. Research indicates that the scale has a sound structural framework, strong item generalizability, and applicability across various contexts. Findings support its reliability and validity as a measure of social support (Shakespeare-Finch & Obst, 2011).
The Patient Health Questionnaire-15 (PHQ-15) | Baseline, Week 4, Month 2, Month 5, and Month 7
  The Patient Health Questionnaire-15 (PHQ-15) will be used to assess the severity of somatization symptoms. In this study, three additional symptoms-stomach pain, palpitations, and limb numbness-are included to provide a more comprehensive evaluation of somatic symptoms. Each item is rated from 0 ("not bothered at all") to 2 ("severely bothered"). Cutoff points are defined as 5 (mild), 10 (moderate), and 15 (severe somatic symptoms). Findings support the PHQ-15 as a simple, self-administered tool with good reliability and validity for screening and monitoring somatization severity in clinical and research settings (Kroenke et al., 2002).
The State Hopelessness Scale | Baseline, Week 4, Month 2, Month 5, and Month 7
  The State Hopelessness Scale will be used to measure the level of hopelessness. This instrument has demonstrated high construct validity and incremental validity (Dunn et al., 2014).
The Chinese version of the Difficulties in Emotion Regulation Scale (DERS) | Baseline, Week 4, Month 2, Month 5, and Month 7
  The Chinese version of the Difficulties in Emotion Regulation Scale (DERS) will be used to assess difficulties in emotional regulation. The total scale shows an internal consistency reliability of 0.89, with subscales ranging from 0.79 to 0.88. The DERS includes six factors: awareness, clarity, goals, impulse, nonacceptance, and strategies, demonstrating good structural validity (Wang et al., 2007)
the catastrophizing subscale of the Cognitive Emotion Regulation Questionnaire (CERQ) | Baseline, Week 4, Month 2, Month 5, and Month 7
  Four items from the catastrophizing subscale of the Cognitive Emotion Regulation Questionnaire (CERQ) will be used to assess individuals' tendencies toward catastrophic thinking about negative events, minimizing response burden (Li & Li, 2019). The CERQ is a widely used self-report measure with good factorial validity and internal consistency (Cronbach's α = 0.75-0.87), and catastrophizing has been found to correlate closely with depression and anxiety symptoms (Garnefski & Kraaij, 2007).
A self-developed Adult Alexithymia Scale | Baseline, Week 4, Month 2, Month 5, and Month 7
  A self-developed Adult Alexithymia Scale will be used, comprising three dimensions: emotional restraint, difficulty identifying emotions, and emotional meaninglessness. Preliminary results suggest good reliability and validity, with psychometric research currently under publication.
A self-developed Adult Irritability Scale | Baseline, Week 4, Month 2, Month 5, and Month 7
  A self-developed Adult Irritability Scale will be employed, which includes four dimensions: impulsive or destructive behavior toward objects, interpersonal aggression, negative self-perception, and aggressive impulses or actions. Studies indicate good reliability and validity, and supporting research is currently under review for publication.
The Family Attitude Scale (FAS) | Baseline, Week 4, Month 2, Month 5, and Month 7
  The Family Attitude Scale (FAS) will be used to assess levels of expressed emotion (EE) within families, particularly expressions of anger, hostility, and criticism. The FAS is a 30-item measure that can be completed by any informant to provide an effective assessment of family climate. Findings show that the FAS has high internal consistency, good inter-rater reliability in assessing anger-related behaviors, and strong predictive validity (Kavanagh et al., 1997).
The Caregiver Strain Questionnaire (CSQ) | Baseline, Month 2, Month 5, and Month 7
  The Caregiver Strain Questionnaire (CSQ) will be used to assess stress experienced by family caregivers of children and adolescents with emotional and behavioral disorders. The scale contains two dimensions: subjective strain and objective strain. Studies have demonstrated that the CSQ possesses good reliability and validity (Brannan et al., 1997).
An adapted version of the Intervention Usability Scale (IUS) | Week 4
  An adapted version of the Intervention Usability Scale (IUS) (Aaron R. Lyon et al., 2021) will be used to assess caregivers' evaluations of the usability of parent-child interaction methods. Usability is defined as the extent to which specific users can achieve goals effectively, efficiently, and satisfactorily within a given context. The IUS total score assesses overall usability of the intervention.
laboratory assessments and peripheral venous blood collection | Baseline, Week 4
  To further explore the mechanisms and potential biological underpinnings of the intervention, laboratory assessments and peripheral venous blood collection will be conducted at baseline and at the end of the intervention (Week 2). Laboratory tests (e.g., blood count and biochemical indicators) will assess general physiological conditions before and after treatment. Peripheral blood samples will be used for genetic analysis to identify potential biomarkers associated with suicide risk and intervention response.
Sheehan Disability Scale (SDS) | Baseline, Week 4, Month 2, Month 5, and Month 7
  The Sheehan Disability Scale (SDS), developed by Sheehan (1983), is a brief self-report instrument designed to assess functional impairment associated with mental disorders, particularly depression and anxiety. The scale measures the extent to which symptoms disrupt an individual's daily functioning across three key domains: work/school performance, social life/leisure activities, and family life/home responsibilities. Each domain is rated on a 0-10 visual analog scale, where 0 indicates "no impairment" and 10 indicates "extreme impairment." The total score, obtained by summing the three items (range: 0-30), reflects the overall level of disability, with higher scores denoting greater functional impairment.
  The SDS is valued for its brevity, ease of administration, and sensitivity to treatment effects. It provides a quick yet robust estimate of functional outcomes complementary to symptom severity scales such as the PHQ-9 or HAM-D.
Clinical Global Impression - Efficacy Index (CGI-E) | Week 4
  The CGI-E evaluates therapeutic efficacy relative to side effects using an NIMH-defined matrix. Higher values indicate greater net clinical benefit.
the Client Satisfaction Questionnaire (CSQ) | Week 4
  After completing the intervention, participants will complete the Client Satisfaction Questionnaire (CSQ), an 8-item self-report measure designed to assess overall satisfaction with the quality, effectiveness, and experience of treatment services. Each item is rated on a 4-point Likert scale, with higher scores indicating greater satisfaction. The questionnaire also includes an open-ended section allowing participants to provide qualitative feedback regarding their treatment experience. Research has demonstrated that the CSQ has good internal consistency and shows strong convergent validity with other satisfaction measures (Attkisson & Greenfield, 2004).
the Working Alliance Inventory (WAI) | Week 4
  At the end of the intervention, participants will complete the Working Alliance Inventory (WAI), a 12-item questionnaire designed to evaluate the therapeutic relationship between the participant and the counselor. Higher total scores indicate a stronger and more positive therapeutic alliance (Gaston, 1991).
an adapted version of the Working Alliance Inventory (WAI) | Week 4
  After the intervention, therapists will complete an adapted version of the Working Alliance Inventory (WAI), consisting of 12 items designed to assess the therapist's perception of the therapeutic relationship with the client. Higher scores indicate a stronger and more effective therapeutic alliance (Gaston, 1991).
CGI-Improvement (CGI-I) | Week 4
  The Clinical Global Impression (CGI) scale, developed by the U.S. National Institute of Mental Health (NIMH) in 1976, is a clinician-rated tool that provides a global assessment of a patient's illness severity, improvement, and therapeutic response. The CGI-I assesses overall change from baseline on a 7-point scale (1 = very much improved, 7 = very much worse).

OTHER OUTCOMES:
The Intervention Usability Scale (IUS) | Week 4
  The Intervention Usability Scale (IUS) (Aaron R. Lyon et al., 2021) will be used to assess therapists' perceptions of the usability of the intervention. Usability is defined as the degree to which a specific user can achieve goals effectively, efficiently, and satisfactorily in a given context. The IUS comprises two dimensions-Usability and Learnability-and demonstrates good internal consistency, with Cronbach's α coefficients of 0.83 (total), 0.84 (usability), and 0.67 (learnability), indicating acceptable reliability.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Sixth Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
The decision on sharing de-identified individual participant data (IPD) has not yet been finalized and will depend on ethical approval, participant consent, and institutional policies at the time of study completion.